CLINICAL TRIAL: NCT01338779
Title: Identification and Mechanistic Investigations of Tolerant Transplant Recipients
Brief Title: Study of Tolerant Kidney Transplant Recipients
Acronym: FACTOR
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN507ST; NCT00083655 (obsolete NCT alias)
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Transplant Rejection; Kidney Transplantation; Renal Transplantation; Renal Transplant; Transplant Tolerance
Keywords: Tolerance; Renal; Allograft; B Cell Signature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine and tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (11):
- Group 1 - kidney tolerant: Renal allograft recipients showing functional tolerance (normal and stable renal function) after discontinuation of immunosuppressive medications for at least 1 year (or based on the investigator's discretion).
- Group 2 - acceptor: Enrollment for group 2 was closed. Renal transplant recipients with functioning allografts (not on dialysis) who had not received immunosuppressive medications for at least 1 year (or at investigator's discretion) but who had moderately impaired or gradually deteriorating renal function, defined as creatinine clearance (CrCl) < 40 mL/min and/or creatinine > 50% above baseline value, and thus did not qualify for group 1.
- Group 3 - kidney graft loss: Enrollment for group 3 is closed. These were renal transplant recipients who had subsequently rejected and lost function of their transplanted kidney.
- Group 4 - kidney monotherapy: Renal transplant recipients showing stable and normal renal function after receiving only prednisone 10 mg/day for at least 1 year (or based on the investigator's discretion).
- Group 5 - kidney standard immunotherapy: Enrollment for group 5 is closed. Stable renal transplant recipients currently on standard immunosuppression.
- Group 6 - kidney chronic rejector: Enrollment for group 6 is closed. Chronic allograft nephropathy group.
- Group 7 - kidney identical twin: Enrollment for group 7 is closed.
- Group 8 - living kidney donors: Corresponding to recipients in group 1 or 4.
- Group 9 - healthy controls: Enrollment for group 9 is closed.
- Group 10 - liver tolerant: Enrollment for group 10 is closed. Liver allograft recipients with functional tolerance (stable and normal liver function) after cessation of immunosuppressive medications for at least three years (or at investigator's discretion).
- Group 11 - liver standard immunotherapy: Enrollment for group 11 is closed. Subjects with a liver transplant who never had an attempt made to discontinue gradually their immunosuppression and who are currently taking standard immunosuppressive medications and have stable and normal liver allograft function after at least 1 year of receiving these drugs.

SUMMARY:
The purpose of this multi-center (observational) registry study is to establish a database of clinical and laboratory information that may help to identify any unique characteristics of tolerant participants that differ from participants who reject their kidney after discontinuing immunosuppressive drugs.

DETAILED DESCRIPTION:
Following kidney (renal) transplantation, one possible complication is rejection of the new kidney. This occurs as a results of the body's immune system attacking (or rejecting) the newly transplanted kidney. After transplant, medicines known as "immunosuppressive" or "anti-rejection" drugs are given to transplant recipients to help prevent rejection of the transplanted kidney. If a transplant recipient stops taking these medicines, they almost always reject their transplanted kidney. However, in some exceptionally rare instances, transplant recipients who stop taking these drugs do not reject their kidney, and the kidney keeps working. The recipients are said at that point to "tolerate" the transplanted kidney, and this condition is referred to as "tolerance".

In this study, participants will be asked to provide consent for the collection of extensive demographic and clinical information; medical histories; and blood and urine samples. Blood and urine samples collected will be used to perform specific assays to help define mechanisms of tolerance.

Originally the study included 11 groups as listed; however, at present only groups 1,4, and 8 remain active. Whereas the initial study duration was 6 years, this was extended to 11 years in order to follow over more extended time a B cell signature identified for tolerant kidney subjects and how this signature may change. (Refer to publications section: Newell, Kirk et al, J Clin Invest. 2010).

ELIGIBILITY:
Inclusion Criteria:

* Must be a renal transplant recipient or living donor
* Meet the criteria for inclusion in one of the study enrollment groups
* Provide informed consent

Exclusion Criteria:

* AIDS [includes all HIV-infected persons who have less than 200 cells/mm(3) CD4+ T-lymphocytes/microL, or a CD4+ T-lymphocyte/micro liter or a CD4+ T-lymphocyte percent of total lymphocytes less than 14, or who have been diagnosed with an AIDS-defining condition as defined by the Centers for Disease Control and Prevention (CDC)
* Current malignancy requiring recent surgery, ongoing chemotherapy or radiation
* Acute systemic infections within 30 days prior to enrollment
* Pregnancy
* Transplant of another organ

Note: Patients meeting any of the exclusion criteria, if identified to have been clinically tolerant prior to the occurrence of the excluding condition, will be enrolled and demographic data collected for the registry; however, the decision as to whether or not to collect blood, urine, and tissue samples will be deferred until the participant's condition improves and the clinically tolerant state persists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Primary Care Clinics
  * Major Kidney (Renal) Transplant Programs
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2004-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To identify individuals who have received a kidney transplant and who have achieved a state of immune tolerance to graft | 0 to 11 years
To create an electronic registry of data on the tolerant and comparison groups that will serve as the basis for statistical analyses | 0 to 11 years
To use data from the registry to perform classical tests of hypotheses regarding the establishment of immune tolerance | 0 to 11 years
To use data from the registry to create and assess predictive statistical models to model such variables as clinical features, duration of tolerant state, and time to onset of immune sensitization | 0 to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Newell, MD, PhD, Study Chair — Emory University
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - NIH Clinical Center, Bethesda, Maryland
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access is available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.

REFERENCES:
- [Background] Schroppel B, Heeger PS. Gazing into a crystal ball to predict kidney transplant outcome. J Clin Invest. 2010 Jun;120(6):1803-6. doi: 10.1172/JCI43286. Epub 2010 May 24. PMID 20501950
- [Result] Newell KA, Asare A, Kirk AD, Gisler TD, Bourcier K, Suthanthiran M, Burlingham WJ, Marks WH, Sanz I, Lechler RI, Hernandez-Fuentes MP, Turka LA, Seyfert-Margolis VL; Immune Tolerance Network ST507 Study Group. Identification of a B cell signature associated with renal transplant tolerance in humans. J Clin Invest. 2010 Jun;120(6):1836-47. doi: 10.1172/JCI39933. Epub 2010 May 24. PMID 20501946
- [Result] Haynes LD, Jankowska-Gan E, Sheka A, Keller MR, Hernandez-Fuentes MP, Lechler RI, Seyfert-Margolis V, Turka LA, Newell KA, Burlingham WJ. Donor-specific indirect pathway analysis reveals a B-cell-independent signature which reflects outcomes in kidney transplant recipients. Am J Transplant. 2012 Mar;12(3):640-8. doi: 10.1111/j.1600-6143.2011.03869.x. Epub 2011 Dec 7. PMID 22151236
- [Result] Newell KA, Asare A, Sanz I, Wei C, Rosenberg A, Gao Z, Kanaparthi S, Asare S, Lim N, Stahly M, Howell M, Knechtle S, Kirk A, Marks WH, Kawai T, Spitzer T, Tolkoff-Rubin N, Sykes M, Sachs DH, Cosimi AB, Burlingham WJ, Phippard D, Turka LA. Longitudinal studies of a B cell-derived signature of tolerance in renal transplant recipients. Am J Transplant. 2015 Nov;15(11):2908-20. doi: 10.1111/ajt.13480. Epub 2015 Oct 13. PMID 26461968
- [Result] Yu J, Steck AK, Babu S, Yu L, Miao D, McFann K, Hutton J, Eisenbarth GS, Klingensmith G. Single nucleotide transcription factor 7-like 2 (TCF7L2) gene polymorphisms in antiislet autoantibody-negative patients at onset of diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):504-10. doi: 10.1210/jc.2007-2694. Epub 2008 Dec 2. PMID 19050058
- [Result] Brennan DC, Shannon MB, Koch MJ, Polonsky KS, Desai N, Shapiro J. Portal vein thrombosis complicating islet transplantation in a recipient with the Factor V Leiden mutation. Transplantation. 2004 Jul 15;78(1):172-3. doi: 10.1097/01.tp.0000128332.71657.ea. No abstract available. PMID 15257060
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: ImmPort Study ID: SDY546 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY546
- Available data/document: Study Protocol: ImmPort Study ID: SDY546 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY546
- Available data/document: Study summary,-design, demographics,mechanistic assays,-study files et al.: ImmPort Study ID: SDY546 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY546
- Available data/document: Individual Participant Data Set: Study ID: FACTOR/ITN507ST — http://www.itntrialshare.org/project/Studies/ITN507STAJT/Study%20Data/begin.view — FACTOR/ITN507ST is the Study Identifier in the ITN TrialShare Clinical Trials Research Portal.
- Available data/document: Original articles w/data and reports; abstracts et al.: Study ID: FACTOR/ITN507ST — http://www.itntrialshare.org/project/Studies/ITN507STAJT/Study%20Data/begin.view — FACTOR/ITN507ST is the Study Identifier in the ITN TrialShare Clinical Trials Research Portal.